CLINICAL TRIAL: NCT01520142
Title: A Two-Part, Randomized, Placebo-Controlled Study to Investigate the Safety, Tolerability and Pharmacodynamic Activity of JNJ-26528398 in Healthy Male Subjects Employing the Intravenous Endotoxin-Induced Model of Acute Inflammation
Brief Title: Safety, Tolerability and Pharmacodynamic Activity of JNJ-26528398 in Healthy Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR100754; 26528398EDI1001 (Other: Janssen Research & Development, LLC); 2011-004459-38 (EudraCT Number)
Record Dates: First submitted 2011-12-09; First posted 2012-01-27 (Estimated); Last update posted 2013-06-24 (Estimated); Status verified 2013-06

CONDITIONS: Healthy Participants
Keywords: Healthy participants; Pharmacodynamic; Pharmacokinetics; Intravenous Endotoxin-Induced Model; Acute Inflammation; JNJ-26528398; Anti-inflammatory

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment (Experimental)
  Interventions: Drug: JNJ-26528398
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: JNJ-26528398 — In Study Part 1, the participant will receive an oral solution of JNJ-26528398 3 mg once daily for 7 days. The same dosing regimen is planned for Part 2, but may be adjusted (lower dose and/or fewer dosing days) based on the data from Part 1.
  Arms: Treatment
Drug: Placebo — In both Study Part 1 and Part 2, the participant will receive an oral solution of matching placebo once daily for up to 7 days.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the anti-inflammatory properties of JNJ-26528398 using an intravenous (IV) endotoxin-induced model of acute, transient inflammation.

DETAILED DESCRIPTION:
This is a 2-part, single center, double-blind study (neither physician nor participant knows the treatment that the participant receives). Part 1 is designed to evaluate the safety, tolerability, and pharmacokinetics (level of drug in the blood) of a dosing regimen of an investigational drug (JNJ-26528398) prior to its use in Part 2. In Part 1, participants will be assigned by chance to receive either 3 mg/day JNJ-26528398 (6 participants) or placebo (3 participants) for 7 consecutive days while staying in the clinic for 10 days. Placebo is an inactive substance that is compared with a drug to test whether the drug has a real effect. Part 2 is designed to evaluate the anti-inflammatory properties of JNJ-26528398 by measuring markers of inflammation in the blood after intravenous (IV) administration of a substance (endotoxin) which activates the immune system and temporarily causes flu-like symptoms. In Part 2, participants will be assigned by chance to receive up to 3 mg/day JNJ-26528398 (6 participants) or placebo (4 participants) for up to 7 consecutive days while staying in the clinic for 10 days. Endotoxin will be given on the last day of study drug administration. Participants will remain in bed for at least 6 hours after endotoxin administration and will be closely monitored by study personnel.

ELIGIBILITY:
Inclusion Criteria:

* Nonsmoker
* Be in good health on the basis of physical examination, medical history, and electrocardiogram (ECG)
* Must have good exercise tolerance
* Have a body mass index of 18-29 kg/m2, inclusive, and body weight between 60 and 85 kg, inclusive
* Have a history of consistent dental hygiene and dental care
* Must adhere to required contraception (subject and partner, if applicable) during the study and for 3 months after study
* Must agree to not donate sperm during the study and for 3 months after study

Exclusion Criteria:

* Is currently enrolled in an investigational study, has recently received an investigational drug (including investigational vaccines), or has donated blood within 3 months
* Has had a vaccination within past 3 months
* Has history of significant drug or alcohol abuse within past 2 years or has a positive drug screen
* Blood donation within past 3 months
* Part 2 only: Has received endotoxin within past 3 months, or has a known allergy or history of significant adverse reaction to endotoxin or its excipients lactose and polyethylene glycol 6000

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2011-11; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
The TNF-α concentrations in plasma (Part 2) | Days 7-8

SECONDARY OUTCOMES:
Other markers of inflammation in blood (Part 2) | Days 7-8
Profile of Mood States (POMS) (Part 2) | Days 1 and 7
  The POMS Standard Form contains 65 items and assesses six dimensions of mood: tension-anxiety, depression-dejection, anger-hostility, vigor-activity, fatigue-inertia, and confusion-bewilderment. Each item is rated by the participant using a 5-point scale ranging from 1 (not at all) to 5 (extremely).
Incidence of adverse events amongst participants (Parts 1 and 2) | Days -1 to 10 and Day 24
Area under the curve (AUC) of JNJ-26528398 (Parts 1 and 2) | Days 1-10
  Blood concentrations sampled at frequent intervals
Maximum plasma concentration (Cmax) of JNJ-26528398 (Parts 1 and 2) | Days 1-10

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC and Development, L.L.C. Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Antwerp, Belgium